CLINICAL TRIAL: NCT01623817
Title: Effectiveness of Vancomycin Loading Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-09-067
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2012-06

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vancomcyin, maintain dose (No Intervention): This arm is received only maintain dose of vancomycin (15mg/kg twice a day or 1g twice a day).
- Vancomycin loading (Experimental): This group is received loading dose 30mg/kg. Subsequent doses of vancomycin are considered standard of care.
  Interventions: Drug: Vancomycin HCL

INTERVENTIONS:
Drug: Vancomycin HCL — Loading dose of 30mg/kg via central or peripheral intravenous infusion during 2 or 3 hours.
  Maintenance dose of vancomycin is 15mg/kg twice a day or 1g twice a day.
  Other Names: The brand name is the Vancomycin hydrochloride.; It is made by Lilly.
  Arms: Vancomycin loading

SUMMARY:
The goal of tish clinical research study is to identify that loading of vancomycin can facilitate rapid attainment of target trough serum vancomycin concentration.

DETAILED DESCRIPTION:
The Study drug

* Vancomycin : a glycopeptide antibiotic, is the first line agent in the treatment of methicillin resistant staphylococcus aureus

Study design : Randomized controlled trials

Study Drug Administration

* If your doctor believes you are eligible, and you agree to take part in this study, you will be randomized to two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Samsung Medical Center MICU and general wards for infectious diseases and hematology division
* Patients with SIRS (systemic inflammatory response syndrome)
* Intravenous vancomycin therapy deemed necessary

Exclusion Criteria:

* Age less than 20 years
* Age more than 75 years
* Current renal insufficiency defined as estimated Glomerular filtration rate < 50mg/min/1.73 m2 by MDRD equation
* History of adverse events to vancomycin 5. Pregnant woman

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time duration for concentration of vancomycin to reach target trough of 15-20 mg/L | Peak level drawn 1 hour after the completion of loading dose. Sequential trough level drawn 30 min before each standard dose for the next 4 doses.

SECONDARY OUTCOMES:
Adverse event rate in each arm, including nephrotoxicity and rash. | 7 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Ran Peck, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea